CLINICAL TRIAL: NCT01286831
Title: An Open-label, Single-arm Study to Determine the Excretionbalance and Metabolic Disposition of [14C]GW642444administered as a Single Dose of an Oral Solution to Healthy Malevolunteers
Brief Title: A Single Dose Study to Determine the Excretion, Balance and Metabolic Disposition of Radiolabelled GW642444.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 106181
Record Dates: First submitted 2010-05-06; First posted 2011-01-31 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Accelerator Mass Spectrometry (AMS); Beta-2 agonist; Absorption, Distribution, Metabolism and Excretion (ADME); Radiolabel
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [14C]GW642444 (Experimental): Single 200μg dose of [14C]GW642444 given on Day 1.
  Interventions: Drug: [14C]GW642444

INTERVENTIONS:
Drug: [14C]GW642444 — Single 200μg dose of [14C]GW642444 given on Day 1.

SUMMARY:
The purpose of this study is to characterise the metabolic disposition of radiolabelled GW642444 when administered orally.

DETAILED DESCRIPTION:
This will be a single-centre, open-label, single-dose study to characterise the metabolic disposition of oral [14C]GW642444. Six healthy male subjects will be enrolled to ensure at least four fully evaluable subjects. Each subject will receive a single 200μg oral dose of GW642444 containing 2 μCi (0.074MBq) of [14C]GW642444. Whilst subjects are inhouse, blood, urine and faecal samples will be collected for a minimum of 168 hours after dosing (7 days) or for up to 240 hours (10 days) depending on amounts of radioactivity still being excreted after Day 5. Faecal sample collection may continue at home for up to 14 days. Bile samples will be collected using Entero-Test string sampling of duodenal bile. Plasma will be prepared from blood at various sample times after dosing to measure parent drug and total radiolabelled drug-related material. Urine and faeces aliquots will be taken to measure total radiolabelled drug-related material. Samples of urine, faeces, plasma and bile will be transferred into a separate study to characterise and, where feasible, quantify metabolites in these matrices. Safety and tolerability will be assessed by blood pressure, heart rate, 12- lead electrocardiogram (ECG), clinical laboratory safety tests, and collection of adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male aged between 30 and 55 years inclusive, at the time of signing the informed consent. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population, which are deemed to be clinically relevant, should always be excluded from enrollment.
2. Body Mass Index (BMI) within the range 18.5-29.0 kg/m2 (inclusive).
3. Subjects who are current non-smokers, who have not used any tobacco products in the 12 month period preceding the screening visit, and have a pack history of ≤ 5 pack years. [number of pack years = (number of cigarettes per day/20) x number of years smoked]
4. AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
5. No significant abnormality on 12-lead ECG at screening. Selected specific ECG findings that are considered to be significant and will exclude the subject from study participation include, but are not limited to, the following:

   * Sinus bradycardia <45bpm
   * Sinus tachycardia ≥110bpm
   * Multifocal atrial tachycardia (wandering atrial pacemaker with rate >100bpm)
   * PR interval >240msec
   * Evidence of Mobitz II second degree or third degree atrioventricular (AV) block.
   * Pathological Q waves (defined as wide [>0.04 seconds] and deep [>0.4mV (4mm with 10mm/mV setting)] or >25% of the height of the corresponding R wave, providing the R wave was >0.5mV [5mm with 10mm/mV setting], appearing in at least two contiguous leads.
   * Evidence of ventricular ectopic couplets, bigeminy, trigeminy or multifocal premature ventricular complexes.
   * QTcF ≥450msec or uncorrected QT >600msec or an ECG that is unsuitable for QT measurements (e.g., poor defined termination of the T wave) Note: QTcF ≥450msec or uncorrected QT >600msec should be confirmed by three readings at least 5 minutes apart.
   * ST-T wave abnormalities (excluding non-specific ST-T wave abnormalities)
   * Right or left complete bundle branch block
   * Clinically significant conduction abnormalities (e.g., left bundle branch block, Wolff-Parkinson-White syndrome)
   * Clinically significant arrhythmias (e.g., atrial fibrillation with rapid ventricular response, ventricular tachycardia)
6. No significant abnormality on the Holter ECG at screening.
7. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:

  1. As a result of medical interview, physical examination or screening investigations, the principal investigator or delegate physician deems the subject unsuitable for the study. Subjects must not have a systolic blood pressure above 145 mmHg or a diastolic pressure above 90 mmHg.
  2. Females.
  3. The subject has been treated for or diagnosed with depression within six months of screening or has a history of significant psychiatric illness.
  4. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
  5. Surgical procedures on digestive tract including corrective surgery for appendicitis (in the 3 months prior to screening) or diverticulitis, cholecystectomy (gallbladder removal), and/or cholelithotomy (gallstone removal).
  6. History of or current spastic/ hyperactive colon.
  7. Subjects who do not have regular defecation patterns (regular defined as passing faeces at least once every two days).
  8. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
  9. Any adverse reaction including immediate or delayed hypersensitivity to any β2-agonist or sympathomimetic drug, or known or suspected sensitivity to the constituents of the GW642444formulation for oral administration.
  10. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
  11. History of alcohol/drug abuse or dependence within 12 months of the study. Abuse of alcohol defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males). One unit is equivalent to a 285mL glass of full strength beer or 425mL schooner of light beer or 1 (30mL) measure of spirits or 1 glass (100mL) of wine (NHMRC Guidelines [NHMRC, 2001]).
  12. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 60 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
  13. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
  14. Participation in a clinical trial involving administration of 14C-labelled compound(s) within the last 12 months. A subjects previous effective dose will be reviewed by the medical investigator to ensure there is no risk of contamination / carryover into the current study.
  15. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
  16. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
  17. The subject has tested positive for HIV antibodies.
  18. A positive urine drug screen at screening, on admission to the unit, or when randomly tested during the study.
  19. Positive alcohol urine test at screening or on admission to the Unit.
  20. Positive urine cotinine test at screening.
  21. Consumption of seville oranges, pomelos (members of the grapefruit family) or grapefruit juice from 7 days prior to the first dose of study medication.
  22. Unwillingness or inability to follow the procedures outlined in the protocol.
  23. Subject is mentally or legally incapacitated.

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2010-05-18 (Actual); Primary Completion 2010-07-09 (Actual); Study Completion 2010-07-09 (Actual)

PRIMARY OUTCOMES:
AUC(0-∞), AUC(0-t), Cmax, tmax, λz and t1/2 of total drug-related material (radioactivity) in plasma following oral dosing. | Two months from first dose.
AUC(0-t), Cmax and tmax of GW642444 following oral dosing. | Two months from first dose.
Urinary and faecal cumulative excretion as a percentage of the total radioactive dose administered over time. | Two months from first dose.

SECONDARY OUTCOMES:
Characterisation of metabolites in plasma, urine, duodenal bile and faecal homogenates. | One year from last subject last visit
Vital signs, 12-lead ECG, Clinical laboratory tests, AEs. | Two weeks from first dose.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Zuidlaren, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Harrell AW, Siederer SK, Bal J, Patel NH, Young GC, Felgate CC, Pearce SJ, Roberts AD, Beaumont C, Emmons AJ, Pereira AI, Kempsford RD. Metabolism and disposition of vilanterol, a long-acting beta(2)-adrenoceptor agonist for inhalation use in humans. Drug Metab Dispos. 2013 Jan;41(1):89-100. doi: 10.1124/dmd.112.048603. Epub 2012 Oct 4. PMID 23043183
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 106181 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/106181?search=study&study_ids=106181#rs
- Available data/document: Study Protocol: 106181 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106181 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106181 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106181 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106181 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106181 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 106181 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register